CLINICAL TRIAL: NCT02413216
Title: Creating a Computerized Self-administered Version of Comprehensive Behavioral Intervention for Tics
Brief Title: TicHelper: A Computerized Comprehensive Behavioral Intervention for Tics (CBIT)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Marquette University (Other)
Responsible Party: Principal Investigator, Mike Himle, Associate Professor, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2R44MH096344-02 (NIH)
Record Dates: First submitted 2015-04-01; First posted 2015-04-09 (Estimated); Last update posted 2017-12-18 (Actual); Status verified 2017-12

CONDITIONS: Tourette's Disorder; Persistent (Chronic) Motor or Vocal Tic Disorder
Keywords: Tic Disorder; Tourette; Motor tic; Vocal tic; Habit reversal training; CBIT; TicHelper; Behavior Therapy
MeSH Terms: conditions — Tourette Syndrome; Bronchiolitis Obliterans Syndrome; Tic Disorders; Tics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TicHelper (Experimental): In this condition, participants will be provided with a secure username and login information for TicHelper.com. Participants will be asked to log in and use TicHelper.com for 8 weeks as instructed by the program (TicHelper recommends 30-60 minutes of website and therapeutic activity per day). TicHelper.com consists of 3 modules: Education, Assessment, and Intervention. The education module provides information about tic disorders and treatment. The assessment module tracks progress through the program. The intervention module uses interactive activities to teach tic management skills including habit reversal training (HRT). During HRT, patients learn to become more aware of tics and pre-tic sensations and to subsequently interrupt tics. Participants will also learn ways to interact with each other regarding tics, to identify and alter tic-worsening factors, and relaxation strategies to reduce stress.
  Interventions: Behavioral: TicHelper
- Internet-Based Resources Condition (Active Comparator): Participants who are assigned to the Internet-Based Resources (IBR) condition will receive a collection of materials with inks to the best available online resources about tic disorders and their treatment. The sites that are provided use a variety of online print, video, and animation materials to teach patients about various aspects of chronic tic disorders and their management. Participants will will be asked to explore and use the website information over the course of 8 weeks in any manner they find helpful. Participants will be asked to spend 30-60 minutes per day reviewing and discussing the information provided.
  Interventions: Other: Internet Based Resources

INTERVENTIONS:
Behavioral: TicHelper — TicHelper.com is an 8-week online program designed to teach tic management skills. Content and activities included in TicHelper.com are based on existing empirically-supported treatments including Habit Reversal Training (HRT) and Comprehensive Behavioral Intervention for Tics (CBIT). TicHelper.com is designed to teach tic management skills including psychoeducation, relaxation training, awareness training, competing response training, and social support. It is also designed to teach patients/parents to recognize and reduce tic-exacerbating reactions and activities.
  Other Names: Habit Reversal Training; Comprehensive Behavioral Intervention for Tics
  Arms: TicHelper
Other: Internet Based Resources — The Internet-Based Resources (IBR) condition is designed to provide patients/parents with access to a wide range of educational materials. These materials contain up-to-date information regarding what is known about tic disorders and their management. Materials covering medical, educational, and behavioral/psychological topics are provided.
  Arms: Internet-Based Resources Condition

SUMMARY:
Tic Disorders (including Tourette Disorder) are relatively common in school-age children and for some children can lead to significant psychosocial and physical impairment and diminished quality of life. Non-pharmacological treatments have been shown to be effective for reducing tics in some children. These treatment options are desired by parents, but are not widely available. The investigators recently developed an online, computerized, self-administered version of CBIT called TicHelper.com. The current study will test the efficacy of TicHelper.com in a randomized clinical trial.

DETAILED DESCRIPTION:
Effective non-pharmacological treatment options such as comprehensive behavioral intervention for tics (CBIT) have been shown to be effective for reducing tics in some children with chronic tic disorders, including Tourette's disorder. Although effective, many parents and children do not have access to a provider trained in these therapies and practical barriers such as travel and high costs for ongoing therapy limit treatment dissemination and utilization.The investigators recently developed an online, computerized, self-administered version of CBIT called TicHelper.com. This program is an 8-week online program designed to teach children and families empirically-supported tic management skills. The current study will test the efficacy of TicHelper.com in a randomized clinical trial in which 64 children with Tourette's Disorder or a persistent (chronic) tic disorder will be randomly assigned to 8-weeks of TicHelper.com (N=32) or an 8-week internet resource control condition (N=32). Tic symptoms will be assessed by a condition-blind independent evaluator at baseline, post-treatment, and 1-month follow-up. Information regarding patient acceptability of the program will also be collected. This project will test whether TicHelper.com is an efficacious and acceptable way to teach tic-management skills for children with tics.

ELIGIBILITY:
Inclusion Criteria:

1. Child and parent are English speaking.
2. Child meets diagnostic criteria for Tourette's disorder or persistent (chronic) motor or vocal tic disorder according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition.
3. Child scores >70 on a brief intelligence test
4. Child currently engages in at least one motor and/or vocal tic multiple times per day
5. Clinician rated tic severity score of > 3 (mildly ill or worse)
6. Child is unmedicated for tics or associated conditions or has been on stable psychotropic medication for at least 6 weeks with no changes or planned changes in dosage.
7. Family has daily access to a personal computer with internet access and software meeting TicHelper minimum system requirements.

Exclusion Criteria:

1. A Yale-Global Tic Severity Scale (YGTSS) score > 30
2. Child scores < 70 on intelligence test
3. Child meets diagnostic criteria for substance abuse or dependence or conduct disorder (within past 3 months) according to the criteria of the Diagnostic and Statistical Manual of Mental Disorders - 5th Edition.
4. Current or past non-drug treatment for tics that consisted of 4 or more sessions of habit reversal training or CBIT.
5. Child has lifetime diagnosis of mania or psychotic disorder
6. Child has any serious psychiatric or neurological condition not currently being managed, managed ineffectively, or requiring more immediate treatment other than that provided by the study.

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 55 (Actual)
Dates: Start 2015-08; Primary Completion 2017-06-01 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Change in the Total Tic Severity Score on the Yale Global Tic Severity Scale (YGTSS) | Baseline, Week 8 (post-treatment), Week 12 (1-month follow-up)
  Clinician interview to assess overall severity of tics

SECONDARY OUTCOMES:
Change in overall tic severity on the Clinician Global Impressions-Severity Scale | Baseline, Week 8 (post-treatment), Week 12 (1-month follow-up)
  Measures clinician's impression of overall severity
Clinician Global Impressions-Improvement Scale | Week 8 (post-treatment)
  Measures clinician's impression of improvement since starting treatment
Clinician Global Impressions- Improvement Scale | Week 12 (1-month follow-up)
  Measures clinician's impression of improvement since starting treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Himle, Ph.D., Principal Investigator — University of Utah; Douglas W Woods, Ph.D., Principal Investigator — Marquette University; Suzanne Mouton-Odum, Ph.D., Principal Investigator — PsycTech, Ltd.
Locations (2):
- United States (2):
  - University of Utah, Salt Lake City, Utah
  - Marquette University, Milwaukee, Wisconsin

REFERENCES:
- [Background] Piacentini J, Woods DW, Scahill L, Wilhelm S, Peterson AL, Chang S, Ginsburg GS, Deckersbach T, Dziura J, Levi-Pearl S, Walkup JT. Behavior therapy for children with Tourette disorder: a randomized controlled trial. JAMA. 2010 May 19;303(19):1929-37. doi: 10.1001/jama.2010.607. PMID 20483969
- [Background] Woods DW, Piacentini JC, Scahill L, Peterson AL, Wilhelm S, Chang S, Deckersbach T, McGuire J, Specht M, Conelea CA, Rozenman M, Dzuria J, Liu H, Levi-Pearl S, Walkup JT. Behavior therapy for tics in children: acute and long-term effects on psychiatric and psychosocial functioning. J Child Neurol. 2011 Jul;26(7):858-65. doi: 10.1177/0883073810397046. Epub 2011 May 9. PMID 21555779
- [Derived] Jakubovski E, Reichert C, Karch A, Buddensiek N, Breuer D, Muller-Vahl K. The ONLINE-TICS Study Protocol: A Randomized Observer-Blind Clinical Trial to Demonstrate the Efficacy and Safety of Internet-Delivered Behavioral Treatment for Adults with Chronic Tic Disorders. Front Psychiatry. 2016 Jun 30;7:119. doi: 10.3389/fpsyt.2016.00119. eCollection 2016. PMID 27445874